CLINICAL TRIAL: NCT03649932
Title: Enteral L Citrulline Supplementation in Preterm Infants - Safety, Efficacy and Dosing
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-0194
Record Dates: First submitted 2018-08-24; First posted 2018-08-28 (Actual); Results first posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-09

CONDITIONS: Bronchopulmonary Dysplasia; Bronchopulmonary Dysplasia Associated Pulmonary Hypertension; Pulmonary Hypertension; Premature Birth; Chronic Lung Disease of Prematurity
Keywords: Bronchopulmonary dysplasia; Pulmonary hypertension; Citrulline
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Hypertension, Pulmonary; Premature Birth

STUDY DESIGN:
Intervention Model Description: Previous studies in patients undergoing cardiac surgery have shown that post-operative pulmonary hypertension did not develop in patients with citrulline level > 37 micromol/L. A cross-sectional study reported that citrulline levels < 29 micromol/L was associated with BPD_PH (100% sensitivity and 75% specificity) hence this may be used as a screening tool for BPD_PH2. The investigators will use the higher levels of citrulline of the reported levels as our goal (>37µmol/L). The investigators will supplement infants with 3 different dosages and check serum levels to see what dose is required to achieve the optimal plasma level of citrulline (>37µmol/L).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- L-citrulline 100 mg/kg/day (Experimental): 50 mg/kg given two times a day (100 mg/kg/day) for total 7 days.
  Interventions: Dietary Supplement: Enteral L-citrulline
- L-citrulline 200 mg/kg/day (Experimental): 100 mg/kg given two times a day (200 mg/kg/day) for total 7 days
  Interventions: Dietary Supplement: Enteral L-citrulline
- L-citrulline 300 mg/kg/day (Experimental): 150 mg/kg given two times a day (300 mg/kg/day) for total 7 days.
  Interventions: Dietary Supplement: Enteral L-citrulline

INTERVENTIONS:
Dietary Supplement: Enteral L-citrulline — L-Citrulline as 10 % solution (100 mg/ml) will be provided to the bedside nurse by the Investigational Pediatric Pharmacy. The drug will be given via gavage feeding by bolus infusions followed by a 0.5 ml water flush twice daily (0900 and 2100). Bolus dosing will be needed due to the small volumes (0.5-1.5 ml per dose in most infants). The volume of nasogastric tubing used in preterm infants (Ameritus 4.0 Fr 50 cm) is 0.48 ml, therefore we will follow the administration with 0.5 ml of saline/water flush to ensure all the study drug is delivered to the patient.
  Administration of study drug - Will be given via gavage feeding tube twice daily (0900 +/- 30 mins, 2100 +/- 30 mins). L-citrulline will be given by the bedside nurse as a bolus followed by 0.5 ml water flush. L-citrulline will be given separate from feeds to avoid any confusion.
  Study drug will be started when infant has been off of TPN for at least 3 days so that IV arginine in TPN does not interfere.

SUMMARY:
Oral L-citrulline supplementation may prevent and/or decrease the severity of chronic lung disease associated with pulmonary hypertension in preterm infants. Since oral L-citrulline supplementation has never been studied in preterm infants before, the side effect profile and appropriate dosing are still unknown. In this pilot study, the investigators will determine the safety profile, efficacy and appropriate dosing of oral L-citrulline in preterm infants. In the future, information from this study will be utilized to conduct a randomized placebo-controlled trial to evaluate the role of L-citrulline supplementation in treating BPD_PH.

DETAILED DESCRIPTION:
Bronchopulmonary dysplasia (BPD) is the most common chronic lung disease in preterm infants (PI). Preterm birth causes disruption in pulmonary vascular growth that leads to decreased vascular surface area that increases pulmonary vascular resistance (PVR). Increased PVR leads to altered vasoreactivity and structural remodeling with intimal hyperplasia and increased muscularization of the small pulmonary arteries. There is no definite treatment for BPD_PH.

Nitric Oxide: Nitric Oxide (NO) is a potent pulmonary vasodilator. Endothelial Nitric oxide synthase (eNOS) mediates production of NO from L-Arginine. L-citrulline is a precursor for L-arginine. L-Arginine is a precursor of nitric oxide (NO). In infants with BPD_PH, there are decreased levels of L-arginine & L-citrulline with decreased production of NO (measured by urinary nitrates & nitrites) leading to increased PVR. Several studies have shown the benefit of oral L-citrulline supplementation in increasing serum citrulline levels, increasing NO production and reducing pulmonary hypertension. Oral L-arginine was not effective in increasing NO production in previous studies and it was due to increased break down of oral L-arginine by intestinal arginases.

Source of L-arginine in preterm infants: Routinely, extremely premature infants receive nutrition as total parental nutrition (TPN i.e. infants get infusion of protein, fat and carbohydrate via central venous line) that contains L-arginine (approximately 1mg/1mL) to metabolize ammonia via urea cycle. PIs receive adequate amount of intra venous arginine from TPN. Routinely, PIs are started with small volumes of enteral feeds which are increased slowly overtime. TPN is slowly decreased as enteral feeds are increasing. As the TPN is going down, intra venous L-arginine intake also drops down and ultimately when the PI are off TPN, they don't get any IV supplemental L-arginine.

Why oral citrulline: Enteral feeds (formula as well as breast milk) is poor source of arginine. Once PIs are on full enteral feed, an enteral feed is the only source of arginine. Interestingly, 40% of enteral arginine gets metabolized by arginase enzyme present in intestine. We speculate that plasma levels of arginine drop once TPN is discontinued and infants are on full feeds. Oral L-arginine has poor bio-availability that is why oral L-arginine supplementation does not increase blood levels of arginine. Since oral citrulline has high bioavailability, the best way to increase serum arginine levels is by oral citrulline supplementation. Oral supplementation of L-citrulline in preterm infants once they are off TPN will likely to increase arginine levels and NO production.

Safety of oral citrulline: L-citrulline has been safely used for decades in patients with urea cycle defects. It has been used in pediatric patients with sickle cell disease and in infants undergoing cardiac surgery. No side effects were reported in these studies. In a study in newborn rats exposed to hyperoxia, L-citrulline caused a marked increase in arginase-2 expression in the lungs and this could have an impact on lung development and remodeling. However, this is only a theoretical risk.

ELIGIBILITY:
Inclusion Criteria:

* Infants less than or equal to 30 weeks' gestational age born at UTMB, Galveston.
* Parents have provided informed consent/assent in a manner that is approved by the IRB

Exclusion Criteria:

* Known congenital or chromosomal anomalies.
* Congenital heart disease affecting cardio-respiratory system (other than PDA, PFO or ASD)
* Necrotizing enterocolitis, sepsis, or any condition requiring surgery prior to recruitment

Max Age: 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amna Investigator, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fike CD, Summar M, Aschner JL. L-citrulline provides a novel strategy for treating chronic pulmonary hypertension in newborn infants. Acta Paediatr. 2014 Oct;103(10):1019-26. doi: 10.1111/apa.12707. Epub 2014 Jun 20. PMID 24862864
- [Background] Montgomery AM, Bazzy-Asaad A, Asnes JD, Bizzarro MJ, Ehrenkranz RA, Weismann CG. Biochemical Screening for Pulmonary Hypertension in Preterm Infants with Bronchopulmonary Dysplasia. Neonatology. 2016;109(3):190-4. doi: 10.1159/000442043. Epub 2016 Jan 19. PMID 26780635
- [Background] Fike CD, Dikalova A, Kaplowitz MR, Cunningham G, Summar M, Aschner JL. Rescue Treatment with L-Citrulline Inhibits Hypoxia-Induced Pulmonary Hypertension in Newborn Pigs. Am J Respir Cell Mol Biol. 2015 Aug;53(2):255-64. doi: 10.1165/rcmb.2014-0351OC. PMID 25536367
- [Background] Vadivel A, Aschner JL, Rey-Parra GJ, Magarik J, Zeng H, Summar M, Eaton F, Thebaud B. L-citrulline attenuates arrested alveolar growth and pulmonary hypertension in oxygen-induced lung injury in newborn rats. Pediatr Res. 2010 Dec;68(6):519-25. doi: 10.1203/PDR.0b013e3181f90278. PMID 20805789
- [Background] Waugh WH, Daeschner CW 3rd, Files BA, McConnell ME, Strandjord SE. Oral citrulline as arginine precursor may be beneficial in sickle cell disease: early phase two results. J Natl Med Assoc. 2001 Oct;93(10):363-71. PMID 11688916
- [Background] Smith HA, Canter JA, Christian KG, Drinkwater DC, Scholl FG, Christman BW, Rice GD, Barr FE, Summar ML. Nitric oxide precursors and congenital heart surgery: a randomized controlled trial of oral citrulline. J Thorac Cardiovasc Surg. 2006 Jul;132(1):58-65. doi: 10.1016/j.jtcvs.2006.02.012. PMID 16798303
- [Background] Abman SH, Hansmann G, Archer SL, Ivy DD, Adatia I, Chung WK, Hanna BD, Rosenzweig EB, Raj JU, Cornfield D, Stenmark KR, Steinhorn R, Thebaud B, Fineman JR, Kuehne T, Feinstein JA, Friedberg MK, Earing M, Barst RJ, Keller RL, Kinsella JP, Mullen M, Deterding R, Kulik T, Mallory G, Humpl T, Wessel DL; American Heart Association Council on Cardiopulmonary, Critical Care, Perioperative and Resuscitation; Council on Clinical Cardiology; Council on Cardiovascular Disease in the Young; Council on Cardiovascular Radiology and Intervention; Council on Cardiovascular Surgery and Anesthesia; and the American Thoracic Society. Pediatric Pulmonary Hypertension: Guidelines From the American Heart Association and American Thoracic Society. Circulation. 2015 Nov 24;132(21):2037-99. doi: 10.1161/CIR.0000000000000329. Epub 2015 Nov 3. PMID 26534956
- [Background] Barr FE, Tirona RG, Taylor MB, Rice G, Arnold J, Cunningham G, Smith HA, Campbell A, Canter JA, Christian KG, Drinkwater DC, Scholl F, Kavanaugh-McHugh A, Summar ML. Pharmacokinetics and safety of intravenously administered citrulline in children undergoing congenital heart surgery: potential therapy for postoperative pulmonary hypertension. J Thorac Cardiovasc Surg. 2007 Aug;134(2):319-26. doi: 10.1016/j.jtcvs.2007.02.043. PMID 17662768
- [Background] Schwedhelm E, Maas R, Freese R, Jung D, Lukacs Z, Jambrecina A, Spickler W, Schulze F, Boger RH. Pharmacokinetic and pharmacodynamic properties of oral L-citrulline and L-arginine: impact on nitric oxide metabolism. Br J Clin Pharmacol. 2008 Jan;65(1):51-9. doi: 10.1111/j.1365-2125.2007.02990.x. Epub 2007 Jul 27. PMID 17662090
- [Derived] Qasim A, Mehdi MQ, Bhatia S, Franco-Fuenmayor ME, Jain SK. Enteral L-citrulline supplementation in preterm infants is safe and effective in increasing plasma arginine and citrulline levels-a pilot randomized trial. J Perinatol. 2024 May;44(5):702-708. doi: 10.1038/s41372-023-01761-x. Epub 2023 Aug 28. PMID 37640809

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose: 50 mg/kg given two times a day (100 mg/kg/day) for total 7 days.
  Enteral L-citrulline: L-Citrulline as 10 % solution (100 mg/ml) will be provided to the bedside nurse by the Investigational Pediatric Pharmacy. The drug will be given via gavage feeding by bolus infusions followed by a 0.5 ml water flush twice daily (0900 and 2100). Bolus dosing will be needed due to the small volumes (0.5-1.5 ml per dose in most infants). The volume of nasogastric tubing used in preterm infants (Ameritus 4.0 Fr 50 cm) is 0.48 ml, therefore we will follow the administration with 0.5 ml of saline/water flush to ensure all the study drug is delivered to the patient.
  Administration of study drug - Will be given via gavage feeding tube twice daily (0900 +/- 30 mins, 2100 +/- 30 mins). L-citrulline will be given by the bedside nurse as a bolus followed by 0.5 ml water flush. L-citrulline will be given separate from feeds to avoid any confusion.
  Study drug will be started when infant has been off of TPN for at least 3 days so that IV arginine in TPN does not interfere.
- Medium Dose: 100 mg/kg given two times a day (200 mg/kg/day) for total 7 days
  Enteral L-citrulline: L-Citrulline as 10 % solution (100 mg/ml) will be provided to the bedside nurse by the Investigational Pediatric Pharmacy. The drug will be given via gavage feeding by bolus infusions followed by a 0.5 ml water flush twice daily (0900 and 2100). Bolus dosing will be needed due to the small volumes (0.5-1.5 ml per dose in most infants). The volume of nasogastric tubing used in preterm infants (Ameritus 4.0 Fr 50 cm) is 0.48 ml, therefore we will follow the administration with 0.5 ml of saline/water flush to ensure all the study drug is delivered to the patient.
  Administration of study drug - Will be given via gavage feeding tube twice daily (0900 +/- 30 mins, 2100 +/- 30 mins). L-citrulline will be given by the bedside nurse as a bolus followed by 0.5 ml water flush. L-citrulline will be given separate from feeds to avoid any confusion.
  Study drug will be started when infant has been off of TPN for at least 3 days so that IV arginine in TPN does not interfere.
- High Dose: 150 mg/kg given two times a day (300 mg/kg/day) for total 7 days.
  Enteral L-citrulline: L-Citrulline as 10 % solution (100 mg/ml) will be provided to the bedside nurse by the Investigational Pediatric Pharmacy. The drug will be given via gavage feeding by bolus infusions followed by a 0.5 ml water flush twice daily (0900 and 2100). Bolus dosing will be needed due to the small volumes (0.5-1.5 ml per dose in most infants). The volume of nasogastric tubing used in preterm infants (Ameritus 4.0 Fr 50 cm) is 0.48 ml, therefore we will follow the administration with 0.5 ml of saline/water flush to ensure all the study drug is delivered to the patient.
  Administration of study drug - Will be given via gavage feeding tube twice daily (0900 +/- 30 mins, 2100 +/- 30 mins). L-citrulline will be given by the bedside nurse as a bolus followed by 0.5 ml water flush. L-citrulline will be given separate from feeds to avoid any confusion.
  Study drug will be started when infant has been off of TPN for at least 3 days so that IV arginine in TPN does not interfere.
Period: Overall Study
Arm/Group | Low Dose | Medium Dose | High Dose
Started | 14 | 14 | 14
Completed | 14 | 13 | 13
Not Completed | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose | Medium Dose | High Dose | Total
Number analyzed (Participants) | 14 | 13 | 13 | 40
Age, Continuous [Median (Standard Deviation); unit: Weeks] | 30 (2.1) | 29.6 (2.5) | 29 (1.5) | 29.4 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 10 | 26
  Male | 6 | 5 | 3 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 6 | 6 | 8 | 20
  African American | 0 | 2 | 0 | 2
  Hispanic | 8 | 5 | 5 | 18
Birth Weight [Median (Standard Deviation); unit: grams] | 1125 (383.5) | 1272 (460) | 1250 (350) | 1250 (393)

OUTCOME MEASURES:

1. Primary Outcome: Change in Plasma Levels of L-arginine and L-citrulline as Measured by LCMS Approach
Description: L-arginine and citrulline levels in the plasma will be measured via liquid chromatography-mass spectroscopy (LCMS) and a change (increase) in plasma levels of 20% on day 7 from baseline on day 0 will be considered significant.
Time Frame: During the week of intervention (day 0 - day 7)
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 14 | 13 | 13
micromol/L
  Citrulline level (day 0) | 24 (9.5) | 33 (17) | 26 (11)
  Citrulline level (day 7) | 112 (85) | 150 (89) | 171 (139)
  Arginine level (day 0) | 56 (63) | 56 (62) | 59 (30)
  Arginine level (day 7) | 91 (63) | 134 (62) | 162 (67)

2. Primary Outcome: Safety of L-citrulline in Preterm Infants: Measured by at Least One Adverse Event
Description: Measured by at least one adverse event that are determined to be related to the study drug.
Time Frame: During the week of intervention (day 0 - day 7)
Measure: Number; unit: Number of Adverse Events
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 14 | 13 | 13
Number of Adverse Events | 0 | 0 | 0

3. Primary Outcome: Number of Participants With an Increase Plasma Level of L-citrulline > 37 Micromol/L
Description: Previous studies have shown that a plasma level of > 37 micromol/L was effective in preventing pulmonary hypertension. This study sought to identify the dosing group of L-citrulline required to increase the plasma level of L-citrulline > 37 micromol/L.
Time Frame: During the week of intervention (day 0 - day 7)
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 10 | 11 | 13
Participants | 8 | 10 | 10

ADVERSE EVENTS:
Time Frame: Adverse event data collected for the week during which study drug was administered.
Arm/Group | Low Dose | Medium Dose | High Dose
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/14 | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-02): https://cdn.clinicaltrials.gov/large-docs/32/NCT03649932/Prot_SAP_000.pdf